CLINICAL TRIAL: NCT03312686
Title: Changes in Esophageal Distensibility With Proton Pump Inhibitors in Patients With Esophageal Eosinophilia: A Pilot Study
Acronym: EOE
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Akira Saito, Assistant Professor of Clinical Medicine, Indiana University
Other Study IDs: EOE-endoflip
Record Dates: First submitted 2017-04-21; First posted 2017-10-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Eosinophilic Esophagitis
Keywords: endoflip
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eosinophilic Esophagitis patients: PPI treatment
  Interventions: Diagnostic Test: endoflip

INTERVENTIONS:
Diagnostic Test: endoflip — Resolution of esophageal eosinophilia by a 2-month course of high dose PPI in patients will lead to improvement in esophageal distensibility, and thus should produce improvement in dysphagia symptoms.

SUMMARY:
This pilot study will explore whether treatment of eosinophilic inflammation in the esophagus is associated with an improved distensibility of the esophagus. Furthermore, previous studies of the esophagus using EndoFlip only measured distensibility of the distal esophagus, specifically the distal esophagus and esophagogastric junction. Eosinophilia in EoE has been demonstrated to affect both upper, middle and lower esophagus. The aim is to measure distensibility both proximal and distal, before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of eosinophilia on esophageal biopsy, defined as a peak count of > 15 eosinophils per high power field (HPF) on light microscopy based on biopsies from at least 2 of the 3 biopsy segments (upper, middle and distal esophagus)

Exclusion Criteria:

1. Secondary causes of esophageal eosinophilia has been excluded, such as eosinophilic GI diseases, celiac disease, Crohn's disease, esophageal infection, hypereosinophilic syndrome, drug hypersensitivity, vasculitis, pemphigus, connective tissue diseases, graft vs. host disease
2. Age < 18 or > 65 years
3. Contraindication for biopsy, such as presence of esophageal varices, coagulopathy
4. History of esophageal surgery, gastric or esophageal malignancy, anatomical abnormality, or major primary motility disorder (such as achalasia)
5. Pregnancy
6. Prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the clinic and endoscopy who are undergoing endoscopy with endoflip
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2016-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Esophageal Distensibility before and after treatment | 2 months
  1. Measure the changes in esophageal distensibility before and after treatment with PPI in patients with esophageal eosinophilia

SECONDARY OUTCOMES:
Change in eosinophilia or the number of eosinophils | 2 months
  4. To correlate changes of esophageal mucosa eosinophilia with changes of lumen distensibility in the different segments of the esophagus

CONTACTS AND LOCATIONS:
Overall Officials: Akiro Saito, MD, Principal Investigator — Indiana University School of Medicine
Locations (2):
- United States (2):
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No